CLINICAL TRIAL: NCT07242027
Title: Lactate-to-albumin, CRP-to-albumin and Procalcitonin-to-albumin Ratios Predict Mortality in Critically Ill Adults: a Retrospective ICU Cohort Study
Brief Title: Use of Lactate-to-Albumin, CRP-to-Albumin, and Procalcitonin-to-Albumin Ratios to Predict Mortality in ICU Patients
Acronym: LAR-CAR-PAR
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Other Study IDs: SUM-SKNIPG-LARCARPAR-ICU-2025
Record Dates: First submitted 2025-09-15; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Respiratory Failure; Cardiac Arrest; Circulatory Failure; Critical Illness; Sudden Cardiac Arrest
Keywords: LAR; CAR; PAR; ICU; mortality; prediction
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency; Heart Arrest; Shock; Critical Illness; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Critically ill adult patients admitted to the ICU who survived hospitalization and were discharged alive.
- Non-Survivors: Critically ill adult patients admitted to the ICU who died during the course of hospitalization.

SUMMARY:
This observational study aims to determine whether three blood test ratios - lactate-to-albumin, CRP-to-albumin, and procalcitonin-to-albumin - can predict in-hospital mortality among critically ill adults. The study includes all adult patients admitted in 2024 to the ICU Ward B at the Silesian Center for Heart Diseases (SCCS) in Zabrze. Researchers will analyze retrospective clinical and laboratory data from electronic medical records, including lab values collected at ICU admission, patient demographics, diagnoses, and outcomes. The biomarker ratios will be manually calculated in Excel and statistically evaluated. The main goal is to assess whether these ratios are associated with patient survival and to identify predictive cut-off values to support early risk stratification in the ICU setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to ICU in 2024
* Availability of data for lactate, CRP, procalcitonin, and albumin

Exclusion Criteria:

* Missing outcome data (e.g. unknown survival status)
* Lack of laboratory parameters necessary for ratio calculation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU. Data collected retrospectively from clinical records (AMMS system).
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 100 days from the date of ICU admission
  All-cause in-hospital mortality among ICU patients during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Acute Medicine, Faculty of Medical Sciences in Zabrze, Medical University of Silesia in Katowice, Poland, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to the retrospective nature of the study and the use of sensitive patient health records. The dataset is not publicly available, and consent for external data sharing was not obtained from participants or their legal representatives.